CLINICAL TRIAL: NCT03252223
Title: Ovarian Function in Women With Polycystic Ovary Syndrome
Brief Title: Ovarian Response to Recombinant Follicle Stimulating Hormone in Women With PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jeffrey Chang, MD, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 170684; P50HD012303 (NIH); K12HD001259 (NIH)
Record Dates: First submitted 2017-08-08; First posted 2017-08-17 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Polycystic Ovary Syndrome; Healthy; Anovulation; Hyperandrogenism
Keywords: polycystic ovary syndrome; anovulation; hyperandrogenism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation; Hyperandrogenism | interventions — Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Women with normal menses (Active Comparator)
  Interventions: Drug: Recombinant Follicle Stimulating Hormone
- Women with Polycystic Ovary Syndrome (Active Comparator)
  Interventions: Drug: Recombinant Follicle Stimulating Hormone

INTERVENTIONS:
Drug: Recombinant Follicle Stimulating Hormone — A modified dose-response study will be done using recombinant FSH (r-FSH), injected sc for 3 days at any one dose. r-FSH will be administered at weight-adjusted doses equivalent to 37.5, 75, and 150 IU based on an average weight of 70 kg, which approximates the weight of the average woman in the United States according to the Centers for Disease Control. Therefore, the actual dose of r-FSH will be 0.53 IU/kg for the 37.5 dose group. Accordingly, r-FSH will be repeated at doses of 1.1 IU/kg and 2.2 IU/kg that are equivalent to 75 and 150 IU for a 70 kg subject. Each FSH stimulation test will be assigned randomly and be separated by an interval of 8 weeks.

SUMMARY:
Women with PCOS suffer from anovulation and, as a result, infertility. Efforts to clinically induce ovulation in these women using follicle stimulating hormone (FSH) administered subcutaneously seemingly requires prolonged administration compared to that of ovulatory women without PCOS. The apparent differing ovarian responsiveness to FSH between PCOS and normal women has not been carefully studied. We propose to address this issue by performing a dose-response study and examine ovarian follicle (estrogen, E2) responses to FSH administered subcutaneously in women with PCOS compared to responses observed in normal women.

DETAILED DESCRIPTION:
In women with polycystic ovary syndrome (PCOS) androgen excess is fundamental to the clinical and physiological alterations of this disorder. In particular, androgen overproduction induces distinctive PCO morphology and appears to influence follicle function. Studies conducted in animals and nonhuman primates have demonstrated that androgens increase follicle number and in small antral follicles enhance granulosa cell (GC) responsiveness to gonadotropin stimulation. However, androgens also have been shown to clearly inhibit GC aromatase activity, and in PCOS follicular fluid, androgen content is abnormally increased. Efforts to reconcile these differences are nonexistent. Moreover, appropriate clinical studies to examine the effects of androgen on follicle health in women are lacking. Excessive androgen exposure in women due to functional tumors or high-dose testosterone treatment in F-M transsexuals has been associated with PCO morphology. Use of androgen therapy to promote follicle growth prior to ovarian hyperstimulation in women undergoing in vitro fertilization has not provided consistent results. However, in these studies GC responses to FSH were not carefully assessed, study populations were exclusively women with previously poor ovarian responses to FSH, and women with PCOS were not included. In fact, there are essentially no clinical studies that have addressed in detail the impact of androgen on follicle function in normal or PCOS women. We hypothesize that androgen facilitates GC responses to FSH in normal women and androgen excess further amplifies follicle growth and function in women with PCOS. We propose to study the effect of increased ovarian androgen on follicle function by increasing intraovarian androgen accumulation using aromatase inhibition followed by FSH stimulation. The experiments in this project are designed to provide insight into whether androgen excess facilitates or interferes with follicle function and ovulation in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects determined to have PCOS based on clinical history of irregular menses and clinical or laboratory evidence of hyperandrogenism and polycystic ovaries on ultrasound OR
* Subjects determined to have a clinical history of regular periods.

Exclusion Criteria:

1. Women with hemoglobin less than 11 gm/dl at screening evaluation
2. Women with untreated thyroid abnormalities
3. Pregnant women or women who are nursing
4. Women with BMI > 37
5. Women with known sensitivity to the agents being used
6. Women with diabetes, or renal, liver, or heart disease
7. Women with any hormonal therapy or metformin for at least 2 months prior to study start.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in granulosa cell function in 24 hours intervals following FSH administration | Serum levels will be assessed daily during each 3 day FSH stimulation test and for five days following the initial FSH administration
  Granulosa function will be assessed using estradiol and inhibin levels
Change in follicle count in following FSH administration | With each dose tested, a pelvic ultrasound will be done before and 3 days after commencing FSH
  Number of ovarian follicles will be assessed by pelvic ultrasound
Change in follicular size in following FSH administration | With each dose tested, a pelvic ultrasound will be done before and 3 days after commencing FSH
  Size of ovarian follicles will be assessed by pelvic ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: R. Jeffrey Chang, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No